CLINICAL TRIAL: NCT02111798
Title: Bupropion-Enhanced CM for Cocaine Dependence
Brief Title: Bupropion-Enhanced Contingency Management (CM) for Cocaine Dependence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00090062; DA034-047 (Other: JHU); R01DA034047 (NIH)
Record Dates: First submitted 2014-03-28; First posted 2014-04-11 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Substance Abuse; Cocaine Dependence
Keywords: substance abuse treatment; cocaine dependence; contingency management; abstinence incentives; medication-enhanced behavioral therapy
MeSH Terms: conditions — Substance-Related Disorders; Cocaine-Related Disorders | interventions — Secondary Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo/Abstinence Initiation (Placebo Comparator): In week 2 participants will randomly assigned to receive twice daily capsules filled with placebo powder. At the end of week 6, participants who did not provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial will be assigned to the Abstinence Initiation incentive arm.
  Interventions: Drug: Placebo; Behavioral: Abstinence Initiation
- Bupropion XL/Abstinence Initiation (Active Comparator): In week 2 participants will randomly assigned to receive bupropion 150mg capsules filled with placebo powder. At the end of week 6, participants who did not provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial will be assigned to the Abstinence Initiation incentive arm.
  Interventions: Drug: Bupropion XL; Behavioral: Abstinence Initiation
- Placebo/Relapse Prevention (Placebo Comparator): In week 2 participants will randomly assigned to receive twice daily capsules filled with placebo powder. At the end of week 6, participants who did provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial will be assigned to the Abstinence Initiation incentive arm.
  Interventions: Drug: Placebo; Behavioral: Relapse Prevention
- Bupropion XL/Relapse Prevention (Active Comparator): In week 2 participants will randomly assigned to receive bupropion 150mg capsules filled with placebo powder. At the end of week 6, participants who did provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial will be assigned to the Abstinence Initiation incentive arm.
  Interventions: Drug: Bupropion XL; Behavioral: Relapse Prevention

INTERVENTIONS:
Drug: Placebo — Participants will be randomly assigned to receive placebo powder in twice-daily capsules at the end of week 2.
  Arms: Placebo/Abstinence Initiation; Placebo/Relapse Prevention
Drug: Bupropion XL — Participants will be randomly assigned to receive bupropion XL 150mg/day in twice-daily capsules at the end of week 2.
  Arms: Bupropion XL/Abstinence Initiation; Bupropion XL/Relapse Prevention
Behavioral: Abstinence Initiation — Participants will provide urine samples thrice weekly during weeks 1-6 of the study. Urine samples will be tested immediately onsite for evidence of recent cocaine exposure. Participants who do not provide 3 urine samples that test negative for cocaine by the end of week 6 will be assigned to an Abstinence Incentive condition.
  Arms: Bupropion XL/Abstinence Initiation; Placebo/Abstinence Initiation
Behavioral: Relapse Prevention — Participants will provide urine samples thrice weekly during weeks 1-6 of the study. Urine samples will be tested immediately onsite for evidence of recent cocaine exposure. Participants who provide 3 urine samples that test negative for cocaine will be promptly assigned to a Relapse Prevention incentive condition.
  Arms: Bupropion XL/Relapse Prevention; Placebo/Relapse Prevention

SUMMARY:
This project will examine effects of bupropion extended release (XL) at a dose of 300mg/day for cocaine abstinence among persons receiving methadone for the treatment of opioid use disorder. Participants also earned financial incentives for providing urine samples that tested negative for cocaine. Bupropion was examined for this purpose because of its previously demonstrated efficacy and safety as well as its pharmacological actions at dopamine systems. Participants were randomly assigned to bupropion XL vs. placebo and received different incentive schedules depending on whether they demonstrated abstinence from cocaine early in the study. Outcomes were tracked over a 6-month time frame and the overarching hypothesis was that bupropion (as compared to placebo) would increase the number of urine samples testing negative for cocaine, independent of whether participants demonstrated abstinence from cocaine early in the study.

DETAILED DESCRIPTION:
The efficacy of behavior therapies may be enhanced by certain medications, particularly those that act on dopaminergic systems. The purpose of this project is to examine effects of bupropion on initiation and maintenance of cocaine abstinence in a population of persons being treated with methadone for the treatment of opioid use disorder who are concurrently using cocaine. Bupropion appears to be the most promising medication for this purpose because of its previously demonstrated efficacy and safety as well as its pharmacological actions at dopamine systems.

Participants will be eligible for inclusion in the study if they are 1) enrolled in methadone maintenance treatment, having previously met the criteria for opioid dependence; 2) between the ages of 18 and 65; 3) provide evidence of cocaine dependence (DSM-IV criteria, self-report, and/or urine tests positive for cocaine during the intake process); and 4) are willing to take study medications and adhere to reporting and data collection schedules.

They will be excluded if they have 1) a history of epilepsy or seizure, including alcohol- or cocaine-related seizure; 2) conditions with increased risk of seizure (e.g. head trauma with loss of consciousness > 30 mins), 3) current use (past 30 days) of antidepressants, antipsychotics, theophyllines, systemic steroids, MAO-A inhibitors, 4) recent use (past 30 days of any medication containing bupropion or budeprion (Wellbutrin®, Zyban®), 5) allergy to bupropion or budeprion, 6) liver enzyme levels greater than 3x upper limit of normal (ULN); 7) uncontrolled diabetes mellitus (glucose > 200mg%); 8) severe psychiatric diagnosis: schizophrenia, psychosis, major depression, mania, current suicidal ideation with plan; cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires; 9) severe renal insufficiency (eGFR < 30 ml/min), 10) pregnant, breast feeding or unwilling to use birth control, 11) medical illness that in the view of the investigators would compromise participation in research, 12) advanced HIV infection requiring HAART 13) current eating disorder (anorexia or bulimia), 14) uncontrolled hypertension with blood pressure ( BP) >140/90.

All participants will be randomly assigned to receive bupropion XL (300mg/day) or placebo. In addition, study participants will also receive an add-on incentive-based intervention depending upon whether they provide 6 consecutive-urine samples that test negative for cocaine. Those who provide 6 consecutive negative urine samples will earn incentives for continuing to provide negative sample (Relapse Prevention group) and those who do not achieve this threshold will earn a different schedule of incentives to promote abstinence (Abstinence Initiation). Our hypothesis is that bupropion as compared to placebo treatment will both enhance the number of urine samples testing negative for cocaine. All participants will be eligible to earn $675 in incentives and cocaine use will be monitored via thrice weekly urine samples collected for a 6 month period.

Overall, this research will provide new and valuable information about the use of bupropion XL to enhance provision of cocaine-negative urine samples in persons independent of their early abstinence behaviors. If hypothesized synergies can be demonstrated, the study will point the way to a significant advance in improved treatment outcomes for this critical group of drug abusers. The proposed study is compelling because it conceptually differentiates the two key clinical issues in treatment of stimulant abusers- abstinence initiation and relapse prevention. It uses a design that efficiently and effectively tests a combined treatment approach for each clinical issue and as well examines cognitive function and reinforcement-based mediators. The research will add to understanding of the interplay between brain reinforcement systems and drug-seeking behavior. Finally, it will make an important contribution to behavioral therapy development by exploring a novel solution to limitations previously noted for CM that include lack of response in some patients and relapse after withdrawal of incentives.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in methadone maintenance
* Meets Diagnostic and Statistical Manual of Mental Disorders, Fifth edition (DSM V) criteria for active cocaine use
* Submits one cocaine positive urine sample within 30 days of study start
* Agrees to study procedures

Exclusion Criteria:

* Healthy and without contra-indications to study medication
* Any history of epilepsy or seizure, including alcohol-, sedative-, or cocaine-related seizure
* Any increased risk of seizure such as serious head trauma with a loss of consciousness of more than an hour duration, brain tumor, or other brain pathology increasing risk of seizure.
* Current eating disorder including anorexia or bulimia
* Current use (last 30 days) of antidepressants, antipsychotics, theophyllines, systemic steroids, monoamine oxidase (MAO-A) inhibitors.
* Recent use (last 30 days) of budeprion, zyban®, wellbutrin®, aplenzin®, or any other medication containing bupropion.
* Allergy to bupropion or budeprion
* Liver enzymes greater than 3x ULN (upper limit of normal)
* Uncontrolled diabetes mellitus, or h/o diabetic coma
* Uncontrolled hypertension with BP > 140/90.
* Current psychiatric diagnosis: schizophrenia, psychosis, major depression, mania, current suicidal ideation as determined by MINI psychiatric interview, cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires
* Severe renal insufficiency (eGFR < 30 ml/min)
* Pregnancy or current breast feeding,
* Medical illness that in the view of the investigators would compromise participation in research, such as uncompensated congestive heart failure, recent history of myocardial infarction (<1year), or urologic conditions that inhibit urine collection.
* Advanced HIV infection requiring the use of HAART (Highly Active Anti-Retroviral Therapy), or with CD4 T cell count < 200/uL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-07; Primary Completion 2020-05 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dunn, Ph.D., MBA, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Behavioral Pharmacology Research Unit, Baltimore, Maryland
  - Institute for Behavioral Resources, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ware OD, Sweeney MM, Cunningham C, Umbricht A, Stitzer M, Dunn KE. Bupropion Slow Release vs Placebo With Adaptive Incentives for Cocaine Use Disorder in Persons Receiving Methadone for Opioid Use Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e232278. doi: 10.1001/jamanetworkopen.2023.2278. PMID 36920397

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Abstinence Initiation: Twice daily capsules filled with placebo powder + participants who did not provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial
- Bupropion XL/Abstinence Initiation: Twice daily capsules filled with bupropion extended release, 150mg (300mg daily) + participants who did not provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial
- Placebo/Relapse Prevention: Twice daily capsules filled with placebo + participants who provided >/=3 consecutive negative urine samples during weeks 1-6 of the trial
- Bupropion XL/Relapse Prevention: Twice daily capsules filled with bupropion extended release, 150mg (300mg daily) + participants who did provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial
Period: Overall Study
Arm/Group | Placebo/Abstinence Initiation | Bupropion XL/Abstinence Initiation | Placebo/Relapse Prevention | Bupropion XL/Relapse Prevention
Started | 31 | 32 | 10 | 10
Completed | 20 | 16 | 10 | 7
Not Completed | 11 | 16 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Bupropion XL/Abstinence Initiation: Twice daily capsules filled with bupropion 150mg + participants who did not provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial
- Placebo/Relapse Prevention: Twice daily capsules filled with placebo powder + participants who did provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial
- Bupropion XL/Relapse Prevention: Twice daily capsules filled with bupropion 150mg + participants who did provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial
- Total: Total of all reporting groups
Arm/Group | Placebo/Abstinence Initiation | Bupropion XL/Abstinence Initiation | Placebo/Relapse Prevention | Bupropion XL/Relapse Prevention | Total
Number analyzed (Participants) | 31 | 32 | 10 | 10 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (4.9) | 46.5 (9.3) | 48.5 (9.8) | 41.3 (11.8) | 45.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 8 | 8 | 23
  Male | 29 | 27 | 2 | 2 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 30 | 31 | 10 | 10 | 81
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 15 | 7 | 6 | 43
  White | 15 | 16 | 2 | 4 | 37
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Cocaine Negative Urines
Description: Comparison of the number of thrice-weekly urine tests submitted during weeks study 7-30 negative for cocaine for persons randomly assigned to receive placebo or bupropion XL during weeks 7-30; excused samples are omitted and missing samples are treated as positive.
Time Frame: Weeks 7-30
Population: Comparisons are conducted as a function of study medication as that is the only variable for which randomization occurred.
Measure: Mean (Standard Error); unit: Mean percent negative urines
Groups:
- Bupropion XL/Abstinence Initiation: Twice daily capsules filled with bupropion XL 150mg + participants who did not provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial
- Bupropion XL/Relapse Prevention: Twice daily capsules filled with bupropion XL 150mg + participants who not provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial
Arm/Group | Placebo/Abstinence Initiation | Bupropion XL/Abstinence Initiation | Placebo/Relapse Prevention | Bupropion XL/Relapse Prevention
Number analyzed (Participants) | 31 | 32 | 10 | 10
Mean percent negative urines | 70.6 (.01) | 57.7 (.01) | 4.2 (.01) | 14.5 (.01)
Statistical Analysis 1: Comparison: Placebo/Abstinence Initiation vs Bupropion XL/Abstinence Initiation vs Placebo/Relapse Prevention vs Bupropion XL/Relapse Prevention; Comparisons were conducted as a function of medication condition, collapsed across abstinence initiation and relapse prevention groups, according to a priori-stated statistical analysis; Test type: Superiority; p = 0.889, Mixed Models Analysis

2. Secondary Outcome: Longest Consecutive Period of Negative Urine Samples
Description: Comparison of the longest string of urine samples testing negative for cocaine that were submitted at thrice weekly visits between weeks 7-30 from persons who were randomly assigned to receive placebo or bupropion XL; samples that were excused are omitted otherwise missing samples are treated as positive.
Time Frame: Weeks 7-30
Measure: Mean (Standard Error); unit: Mean consecutive negative urines
Groups:
- Bupropion XL/Relapse Prevention: Twice daily capsules filled with bupropion Xl 150mg + participants who did provide >/=3 consecutive negative urine samples during weeks 1-6 of the trial
Arm/Group | Placebo/Abstinence Initiation | Bupropion XL/Abstinence Initiation | Placebo/Relapse Prevention | Bupropion XL/Relapse Prevention
Number analyzed (Participants) | 31 | 32 | 10 | 10
Mean consecutive negative urines | 7.8 (2.0) | 11.25 (3.3) | 52.9 (7.0) | 33.3 (7.2)
Statistical Analysis 1: Comparison: Placebo/Abstinence Initiation vs Bupropion XL/Abstinence Initiation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.605, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events represent all events rated as "possibly, probably, or definitely" related to study participation, that were reported by participants to study staff during thrice weekly visits over a 23 week period during study weeks 7 - 30.
Arm/Group | Placebo/Abstinence Initiation | Bupropion XL/Abstinence Initiation | Placebo/Relapse Prevention | Bupropion XL/Relapse Prevention
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/31 | 17/32 | 2/10 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Abstinence Initiation (N=31) | Bupropion XL/Abstinence Initiation (N=32) | Placebo/Relapse Prevention (N=10) | Bupropion XL/Relapse Prevention (N=10)
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Cramps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastro Esophageal Reflux Disease (GERD) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain, Lower Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT02111798/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02111798/ICF_001.pdf